CLINICAL TRIAL: NCT04357964
Title: Beige Fat, Energy, and the Natriuretic Peptide System (ENDA-025-17S)
Brief Title: Beige Fat, Energy, and the Natriuretic Peptide System
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ENDA-025-17S-1; 1IK2CX001678 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: adipose tissue; beige adipose tissue; cardiovascular physiology; B-type natriuretic peptide; metabolism; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and fat biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- obese and lean individuals: obese and lean individuals

SUMMARY:
Obese individuals experience an increased risk of cardiovascular and metabolic diseases. Evidence from genetic studies indicate that the natriuretic peptide (NP) system may protect against these diseases. NP levels differ by obesity status and race has not been established in humans. Thus, the investigators propose a study in which will quantify adipose tissue gene expression and energy expenditure in states of NP deficiency in humans. The overarching postulate is that obese and black individuals have NP deficiencies that contribute to less beige adipose tissue and lower energy expenditure.

DETAILED DESCRIPTION:
Obesity represents a serious public health burden. Obese individuals experience increased risk of cardiovascular and metabolic cardiometabolic disease, including insulin diabetes, resistance, hypertension, and dyslipidemia. Obesity and obesity-associated cardiometabolic dysfunction are significant contributors to morbidity and mortality in Veterans. This indicates that obesity and cardiometabolic dysfunction are complex and multifactorial, and suggests that there are additional factors that contribute to the pathogenesis of obesity and its associated cardiometabolic risk that have been discovered. Moreover, some of the pharmacologic therapies for obesity can have adverse cardiovascular effects. Thus, it is crucial to improve the understanding of the multiple pathways contributing to the pathogenesis of obesity and obesity-associated cardiometabolic risk, including the identification of novel relevant pathways, in order to develop more effective treatments for these diseases. The proposed work will form a foundation for future high-impact studies of mechanisms for adiposity and cardiometabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-55 years
* Body Mass Index (BMI) >= 18.5 and <25 kg/m2 (lean), or BMI 30 kg/m2 (obese)

Exclusion Criteria:

* Significant pulmonary, liver, or renal disease
* Heart failure (any type) or unstable coronary artery disease
* Diabetes Mellitus (Types 1 and 2)
* Thyroid dysfunction
* Active malignancy
* Chronic inflammatory diseases, such as inflammatory bowel disease, hepatitis, rheumatoid arthritis
* Current use of medications likely to affect energy homeostasis, including glucocorticoids, amphetamines, and beta blockers
* Currently pregnant or breastfeeding, or unwilling to avoid becoming pregnant or breastfeeding during study duration
* Significant claustrophobia that would prevent the use of the metabolic cart as part of the study protocol
* Hemoglobin A1c (HbA1c) >= 6.5%
* Liver Function Tests (LFTs) elevated >3x upper limit of normal
* Estimated Glomerular Filtration Rate (eGFR) <40 ml/min
* Currently abnormal thyroid stimulating hormone (TSH)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers who are U.S. veterans
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (2):
- United States (2):
  - VA TVHS Nashville, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled subjects underwent a screening visit to determine eligibility for the study. The screening visit included a medical history, physical examination, calculation of BMI, and a blood draw for CMP, CBC, HbA1c, TSH, and free T4. A pregnancy test was completed on female subjects of child-bearing potential. Eligible subjects who still wished to participate in the study were then enrolled for the main study visit.
Groups:
- Lean Individuals: Body Mass Index (BMI) ≥18.5 and <25 kg/m2 (As defined per protocol)
- Obese Individuals: BMI ≥30 kg/m2 (as defined by protocol)
Period: Overall Study
Arm/Group | Lean Individuals | Obese Individuals
Started | 55 (55 lean participants (all U.S. veterans)) | 82 (82 obese participants (22 obese Veterans, 60 obese individuals from prior study))
Completed (Number of participants analyzed) | 37 (37 lean participants (all U.S. veterans) with complete primary endpoint data (adipose UCP1 gene expression)) | 81 (81 obese participants (21 obese Veterans, 60 obese individuals from prior study) with complete primary endpoint data)
Not Completed | 18 | 1
Not completed — Deemed not to have enough sufficient adipose tissue to undergo subcutaneous adipose biopsy | 5 | 0
Not completed — Did not have usable primary endpoint data due to insufficient or low-quality adipose sample | 13 | 0
Not completed — Adipose sample was insufficient quality | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lean Individuals: lean individuals (BMI >= 18.5 and <25 kg/m2)
- Obese Individuals: obese individuals (BMI>= 30 kg/m2)
- Total: Total of all reporting groups
Arm/Group | Lean Individuals | Obese Individuals | Total
Number analyzed (Participants) | 37 | 81 | 118
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [31.5 to 48] | 52 [41.0 to 57.0] | 47 [37.5 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 50 | 61
  Male | 26 | 31 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 14 | 19
  White | 31 | 64 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 81 | 118

OUTCOME MEASURES:

1. Primary Outcome: Adipose Tissue Gene Expression of UCP1 (Uncoupling Protein 1)- Differences by Obesity Status
Description: Primary endpoint is adipose tissue gene expression of UCP1 (Uncoupling Protein 1)- differences by obesity status (obese vs. lean). Units for primary endpoint are relative UCP1 gene expression (quantified using quantitative real-time reverse-transcription polymerase chain reaction (qRT-PCR)), normalized to a housekeeping gene.
Time Frame: Study Day 1
Population: All participants who had data for primary endpoint (adipose tissue UCP1 gene expression).
Measure: Median (Inter-Quartile Range); unit: fold change
Groups:
- Lean Individuals: lean individuals (BMI between 18.5 and 24.9 kg/m2)
Arm/Group | Lean Individuals | Obese Individuals
Number analyzed (Participants) | 37 | 81
fold change | 7.79 [3.26 to 16.33] | 24.33 [16.5 to 40.93]
Statistical Analysis 1: Comparison: Lean Individuals vs Obese Individuals; Test type: Equivalence — Statistical significance was defined as p< 0.05 for determining difference between groups at baseline in this observational study. There was no treatment intervention in this study, so there is no true equivalence margin; p < 0.01, Kruskal-Wallis — Statistical significance was defined as p< 0.05

2. Secondary Outcome: Associations of Adipose Tissue Gene Expression of UCP1 (Uncoupling Protein 1) With Natriuretic Peptide Markers
Description: The investigators will determine associations of adipose tissue gene expression of UCP1 with natriuretic peptide markers (natriuretic peptide receptor gene expression in adipose tissue, and circulating natriuretic peptide levels)
Time Frame: Study Day 1
Population: Correlation between UCP1 gene expression and natriuretic peptide receptor-C (NPR-C) gene expression. The groups are combined in this analysis because the investigators had pre-specified that this secondary outcome would analyze this correlation across all individuals (lean and obese combined) for whom gene expression data was available.
Measure: Number; unit: correlation coefficient
Groups:
- Obese and Lean Individuals: correlation between UCP1 gene expression and natriuretic peptide receptor-C (NPR-C) gene expression across all individuals
Arm/Group | Obese and Lean Individuals
Number analyzed (Participants) | 118
correlation coefficient | 0.28
Statistical Analysis 1: Comparison: Obese and Lean Individuals; Test type: Equivalence — Statistical significance was defined as p < 0.05. There was no intervention in this study, so there is no true equivalence margin; p < 0.01, Pearson correlation

3. Secondary Outcome: Adipose Tissue Gene Expression of UCP1 (Uncoupling Protein 1)- Differences by Race
Description: The investigators will determine adipose tissue gene expression of UCP1 (Uncoupling Protein 1), and analyze differences by race (blacks compared with whites).
Time Frame: Study Day 1
Population: All participants who had data for primary endpoint (adipose tissue UCP1 gene expression), and who also self-reported their race as "white" or "black".
Measure: Median (Inter-Quartile Range); unit: fold change
Groups:
- Race: Blacks: Race: blacks
- Race: Whites: Race: whites
Arm/Group | Race: Blacks | Race: Whites
Number analyzed (Participants) | 19 | 96
fold change | 14.7 [11.2 to 28.5] | 20.9 [10.0 to 37.3]
Statistical Analysis 1: Comparison: Race: Blacks vs Race: Whites; Test type: Equivalence — Statistical significance was defined as p< 0.05 for determining difference between groups in this observational study. There was no treatment intervention in this study, so there is no true equivalence margin; p = 0.52, Kruskal-Wallis — Statistical significance was defined as p< 0.05

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Description: A total of 22 obese individuals underwent procedures in the current study and thus there were 22 obese individuals "at risk" for an AE in the present study. Separately, we analyzed the baseline samples/data from 60 obese individuals from a previously conducted study, but these subjects were not "at risk" for an adverse event in the present study since they did not undergo procedures in the present study. AE's from this previous study are listed at: https://clinicaltrials.gov/study/NCT03101930.
Groups:
- Lean Individuals: BMI ≥18.5 and <25 kg/m2 (as defined by protocol)
- Obese Individuals: BMI ≥30 kg/m2 (as defined by protocol)
  A total of 22 obese individuals underwent procedures in the current study and thus there were 22 obese individuals "at risk" for an adverse event in the present study. Separately, we analyzed the samples/data from 60 obese individuals from a previously conducted study, but these subjects were not "at risk" for an adverse event in the present study since they did not undergo procedures in the present study.
Arm/Group | Lean Individuals | Obese Individuals
All-Cause Mortality (participants affected / at risk) | 8/55 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/22
Other Adverse Events (participants affected / at risk) | 8/55 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lean Individuals (N=55) | Obese Individuals (N=22)
Local skin reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — Redness, bruising or tenderness around biopsy site.
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Experience nausea during the biopsy procedure.
Lightheaded (Vascular disorders) | 3 (3) | 0 (0) — Experienced lightheadedness during biopsy procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04357964/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT04357964/ICF_000.pdf